CLINICAL TRIAL: NCT05431283
Title: Efficacia Nel Mondo Reale di Tofacitinib Sulla Spondiloartropatia Associata Alla Colite Ulcerosa
Brief Title: Real-world Effectiveness of Tofacitinib on Ulcerative Colitis Associated Spondyloarthropathy
Acronym: RETUCAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Italian Group for the study of Inflammatory Bowel Disease (IG-IBD) (Other)
Responsible Party: Sponsor
Other Study IDs: 007
Record Dates: First submitted 2022-04-06; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Ulcerative Colitis; Spondyloarthropathy
MeSH Terms: conditions — Colitis, Ulcerative; Spondylarthropathies | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tofacitinib — This study aims to assess the effectiveness of TOFA

SUMMARY:
Tofacitinib (TOFA) is a JAK inhibitor already used in rheumatology for the treatment of moderate-to-severe active rheumatoid arthritis and psoriatic arthritis in adult patients who have responded inadequately to, or who are intolerant to one or more disease- modifying antirheumatic drugs. Furthermore, TOFA has been recently approved for the treatment of adult patients with moderate-to-severe active Ulcerative Colitis (UC) who had no response, lose response, or were intolerant to either conventional therapy or a biologic agent. The approval was based on the efficacy demonstrated by TOFA in three phase 3 randomized controlled trials named OCTAVE: two identically designed, 8-week, placebo- controlled, induction studies of oral TOFA 10 mg twice daily followed by the OCTAVE Sustain 52-week maintenance study. About sacroiliitis, 2 out of 8 patients treated with TOFA improved after 8 weeks, compared with 0 out of 3 patients in the placebo group. Obviously, these data should be interpreted with extreme caution since patient numbers were very low, and it should be again emphasized that these trials were not designed to explore the efficacy of TOFA onextraintestinal manifestations.

On these premises, we designed a prospective, multicenter, observational, 52-week study with the aim of assess the effectiveness of TOFA on UC-associated spondyloarthropathy.

DETAILED DESCRIPTION:
Participants will receive TOFA at study entry (week 0) as treatment for UC according to standard clinical practice and recommended dosage of the drug, and will be followed up to 52 weeks. At baseline, all enrolled patients will undergo a detailed assessment including gender, age, duration of disease, smoking status, extension of disease (according to Montreal classification), clinical activity (assessed with the partial Mayo Score), C-Reactive Protein (CRP) values, faecal calprotectin, previous and concomitant therapies, data on SpA (axial vs. peripheral SpA, and assessment of ASDAS-CRP and/or DAS28-CRP scores). The joint response (JR), steroid free joint response (SFJR), clinical intestinal response (CIR), steroid free clinical intestinal remission (SFCIR), CRP and calprotectin values will be assessed at 8, 24 and 52 weeks (see further for the definitions of the outcomes). The burden of UC and therapy with TOFA on work productivity and health- related quality of life will be evaluated through the administration of the Work Productivity and Activity Impairment (WPAI) Questionnaire and the Short Inflammatory Bowel Disease Questionnaire Score (Short IBDQ), respectively, at baseline and at 24 and 52 weeks. The patients will be assessed with direct visits and biochemical evaluations, including monitoring of serum lipid levels, according to the routine clinical practice established for subjects treated with TOFA. The support by a rheumatologist is suggested in the clinical evaluation of patients All data will be collected anonymously in a specifically arranged eCRF form inside the IG-IBD registry.

ELIGIBILITY:
Inclusion Criteria:

* An established diagnosis of UC and an established diagnosis of axial and/or peripheral SpA according to the Assessment of Spondyloarthritis international Society (ASAS) criteria
* Indication for treatment with TOFA as a therapy for UC according to the clinical practice and summary of product characteristics
* Active SpA at baseline assessed with an Ankylosing Spondylitis Disease Activity Score (ASDAS)-CRP ≥ 1.3 in case of axial SpA, and with a disease activity score (DAS)28-CRP ≥ 2.6 in case of peripheral SpA.
* Capability to express a written informed consent for the study

Exclusion Criteria:

Rheumatologic diseases other than UC-associated SpA (for example, previous diagnosis of rheumatoid arthritis or psoriatic arthritis)

* Inactive SpA at baseline
* Inability to understand or sign the informed consent
* Contraindications to treatment with TOFA (pregnancy, risk factors for venous thromboembolism, active infections, hepatic failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 years or older admitted at each IG-IBD center that agrees to participate could be be screened for inclusion
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
joint response and steroid free joint response | week 8
  evaluate the rate of patients achieving joint response and steroid free joint response on Ulcerative Colitis-associated spondyloarthropathy at week 8, 24, and 52
joint response and steroid free joint response | week 24
  evaluate the rate of patients achieving joint response on Ulcerative Colitis-associated spondyloarthropathy
joint response and steroid free joint response | week 52
  evaluate the rate of patients achieving joint response and steroid free joint response on Ulcerative Colitis-associated spondyloarthropathy

SECONDARY OUTCOMES:
clinical intestinal response CIR | week 8
  To assess the rate of patients achieving a clinical intestinal response CIR for Ulcerative Colitis
clinical intestinal response CIR | week 24
  To assess the rate of patients achieving a clinical intestinal response CIR for Ulcerative Colitis
clinical intestinal response CIR | week 52
  To assess the rate of patients achieving a clinical intestinal response CIR for Ulcerative Colitis
steroid free clinical intestinal remission | week 52
  To assess the rate of patients achieving a steroid free clinical intestinal remission for Ulcerative Colitis
impact of Ulcerative Colitis | week 8
  To assess the impact of Ulcerative Colitis and therapy with TOFA on Work Productivity and Activity Impairment through the administration of WPAI Questionnaire at baseline
impact of Ulcerative Colitis | week 24
  To assess the impact of Ulcerative Colitis and therapy with TOFA on Work Productivity and Activity Impairment through the administration of WPAI Questionnaire at baseline
impact of Ulcerative Colitis | week 52
  To assess the impact of Ulcerative Colitis and therapy with TOFA on Work Productivity and Activity Impairment through the administration of WPAI Questionnaire at baseline
health-related quality of life | week 24 and 52
  To assess the health-related quality of life of the patients with the administration of the Short IBDQ at baseline
health-related quality of life | week 52
  To assess the health-related quality of life of the patients with the administration of the Short IBDQ at baseline
adverse events | 24 month
  To report the rate of adverse events with TOFA
redictors of joint response JR, steroid free joint response SFJR, clinical intestinal response CIR, and steroid free clinical intestinal remission SFCIR | 24 month
  To assess the predictors of joint response JR, steroid free joint response SFJR, clinical intestinal response CIR, and steroid free clinical intestinal remission SFCIR

CONTACTS AND LOCATIONS:
Locations (1):
- IBD Unit, Department of Internal Medicine, "Villa Sofia-Cervello" Hospital, Palermo, Italy